CLINICAL TRIAL: NCT02159274
Title: Shoulder Disability and Late Symptoms Following Oncoplastic Breast Surgery
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Danish Cancer Society (Other)
Responsible Party: Sponsor
Other Study IDs: KRH-2014; 1-10-72-335-13 (Other: Research Ethics Committee for Central Region Denmark); 2007-58-0010 (Other: Data tilsynet)
Record Dates: First submitted 2014-06-02; First posted 2014-06-09 (Estimated); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Breast Cancer; Carcinoma in Situ of the Breast
Keywords: Late symptoms; Shoulder function; Cosmetic results; EORTC; Lymphoedema
MeSH Terms: conditions — Breast Neoplasms; Breast Carcinoma In Situ; Lymphedema

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- BCS without oncoplastic techniques: BCS without oncoplastic techniques
- BCS with oncoplastic techniques: BCS with oncoplastic techniques.

SUMMARY:
Breast cancer affects a large proportion of Danish women and late morbidity following breast cancer treatment including pain, reduced motility and force of the arm and shoulder, disturbed sensitivity, and lymph edema affects many patients. The risk for such late complications have previously been carefully described by us and others in patients operated by traditional methods, but the follow-up in most of these studies have been rather short , and long time follow-up results are not available. The impact of the new oncoplastic techniques that allows more women to have breast conserving surgery is not known yet. These operations are more extensive and therefore might be accompanied by more complications. The purpose of this study is to give answer to that question.The study includes three parts. First a questionnaire to patients who have breast conserving surgery performed in one of the three breast units in Central Region Denmark. It contains questions regarding arm morbidity, quality of life, comorbidity, and body image. The questionnaire should be filled in preoperatively and 18 months after surgery. The second part consists of an objective evaluation of shoulder and arm function and cosmesis before and after breast conserving surgery with and without oncoplastic techniques. This should be performed at baseline before surgery and 18 months later. The third part is a long time follow-up of patients after breast conserving surgery without oncoplastic techniques. This group of patients is recruited from three breast units in Central Region Denmark. It contains questions regarding arm morbidity, quality of life, comorbidity, and body image. The questionnaire should be filled in preoperatively and 18 months after surgery. The second part consists of an objective evaluation of shoulder and arm function and cosmesis before and after breast conserving surgery with and without oncoplastic techniques. This should be performed at baseline before surgery and 18 months later. The third part is a long time follow-up of patients after breast conserving surgery without oncoplastic techniques. This group of patients is recruited from the cohort in a previous study with 18 months follow-up following breast conserving surgery without oncoplastic technique.

DETAILED DESCRIPTION:
Aims and perspectives:

During the last 20 years there has been increasing focus on the morbidity following breast cancer treatment. This has lead to new and less mutilating surgical techniques to replace the traditional operations: Breast conserving surgery (BCS) instead of mastectomy and sentinel lymph node dissection (SLND) instead of axillary lymph node dissection (ALND). Lately, oncoplastic techniques have been introduced. These techniques further increase the ability to preserve the breast in breast cancer and are expected to increase the cosmetic results compared with traditional techniques, but they are somewhat larger procedures and might therefore lead to increased morbidity after treatment. Hitherto this has not been evaluated in clinical research trials.

The aim of the present study is to examine if oncoplastic techniques in relation to breast cancer treatment have an independent influence on morbidity and quality of life compared to traditional BCS.

In addition, a group of breast cancer patients treated with BCS 10 years ago and who underwent a similar study back then, will be invited to a reevaluation of shoulder function and morbidity.

Background:

Previously, mastectomy was the most applied surgical procedure related to breast cancer. Until the beginning of 1990's it was, by DBCG (Danish Breast Cancer Cooperative Group), recommended as a standard treatment. During the transition towards a more gentle surgical procedure, the use of oncoplastic techniques has been incorporated1,2.

The definition of oncoplastic breast surgery is defined by DBCG as: "a breast conserving procedure, including techniques of plastic surgery, where traditional breast conserving surgery would have lead to a cosmetic unsatisfactory result, and mastectomy would have been the alternative. The requirement for classifying a procedure as oncoplastic is 'the transfer of tissue that requires further skin incision than the breast conserving surgery in its own'3.

The oncoplastic techniques in breast cancer surgery are divided into 3 groups: volume displacement, volume reduction and volume replacement3-5. The oncological results of oncoplastic breast surgery has been evaluated in other studies and found comparable to the oncological results of traditional BCS and mastectomy6.

Increasing evidence have shown that among breast cancer patients a substantial fraction suffer from late symptoms including impairment of shoulder function, pain, disturbance in sensibility, and lymph edema7-9. The sequels are attributable to treatment related factors, including the breast surgical procedure10, axillary dissection11, and radiation therapy12. Studies indicate that sentinel lymph node biopsy (SNLB) reduces shoulder morbidity as compared to ALND11,13, but shoulder impairment also occur after this procedure14.

Recently, the occurrence of late symptoms has been addressed in two Danish publications based on questionnaires7,8 with 2-3 years8 and more than 5 years7 observation, respectively. These studies showed that chronic pain 2-3 years after surgery is a problem in up to 47% of patients of whom 13% suffered from severe and 39% from moderate pain8. More than five years after treatment, chronic pain was recorded in 29% of patients7, and this was associated with poorer quality of life and a higher medicine consumption. Furthermore, a large part of long time survivors reported arm swelling (25%), phantom symptoms (19%), paresthesia (47%), and allodynia (15%)7.

The reported frequency of Lymph oedema following breast cancer treatment vary considerably, probably depending on different definitions and different methods for measurement. As stated earlier, many patients report a subjective feeling of swelling, though the proportion of affected patients seems lower in studies, where objective measures are applied. In a study on node negative patients comparing the results of sentinel node biopsy (SNB) with axillary dissection (ALND)11 up to 18 months after surgery, arm swelling was reported in 7% and 44%, respectively, emphasizing the advantage of the more limited procedure. Using the water displacement method the difference in arm volume between these groups was very modest, although statistically significant. At 18 months, the arm volume on the operated side was 10 ml less than on the non-affected arm in the SNB group, compared with an increase of 28 ml in the ALND group. The water displacement method has been simplified and validated since15,16.

Shoulder morbidity median three years after surgery including ALND was measured in a study on 132 patients (mastectomy 67%, BCT 33%)10. The shoulder function was assessed by the Constant Shoulder Score (CSS), combining subjective symptoms with objective measures of range of motion (ROM) and strengths. Thirty-five percent of the patients had reductions in ROM, in most cases it was flexion and abduction that were most affected. Among these patients CSS was reduced by 12% on the treated side compared with the non-treated shoulder. Patients with normal ROM had comparable CSS on the two sides. In comparison with BCS and radiotherapy, mastectomy combined with postoperative radiation, more often lead to reduced ROM (OR 8.5). In the study by Husted Madsen et al.11 on more recently operated node negative patients, ALND turned out to be significantly associated with a poorer outcome when the dependent variable was the absence or presence of subjective arm and shoulder complaints.

Most studies concerning morbidity, especially those with objective evaluation of patients, have a short follow-up period typically only a few years. No such studies with long-term follow-up up to 5-10 years are available.

A few studies have aimed at describing the effect of physiotherapy on shoulder-arm morbidity13,17, and they have confirmed a better outcome after physiotherapy including general advice and recommendations about how to use and protect the affected arm and instructions for exercises. In the randomized study by Lauridsen et al.13, team instructed physiotherapy consisting of 12 sessions of 60 minutes twice a week instituted between the 6th and 8th postoperative week was compared to the same treatment postponed until the 26th postoperative week. The team instructed physiotherapy commenced early immediately improved the shoulder function, but the same treatment could improve shoulder function significantly even when instituted as long as six months postoperatively.

In a recently published randomized study, Veiga et al.18 have found indications of a better quality of life and self-esteem in BCS including oncoplastic surgery than in patients undergoing traditional BCS. On the other hand, in a study including 101 patients it was found that breast symmetry after BCS had had no effect on quality of life19. In that study symmetry was evaluated by a breast analyzing tool (BAT), one of more available objective measures. Most often, symmetry has been evaluated subjectively by a panel of experts, which has been considered the gold standard. Lately, Cardoso et al. have introduced another objective method where the cosmetic outcome is evaluated semi-automatically from systematic clinical fotos20. They reported a 70% agreement between the expert panel and their measurements. The cosmetic outcome after BCS has been evaluated by Lyngholm et al.21 using the "breast retraction assessment" (BAT) which estimates the symmetry based on measurements on clinical photos22.

The relation between the oncoplastic surgical techniques and shoulder disability, chronic pain, and lymph edema has hitherto not been systematically investigated, but some attempts have been made to describe the impact on shoulder function of post-mastectomy reconstructive surgery. In a study from Sweden23, shoulder function after reconstructive procedures involving the latissimus dorsi flap was examined. The main finding was that the reconstruction lead to an insignificant increase in long-term shoulder morbidity, but it was also noted that a small subset of patients developed long-term impairment.

Design and methods:

The study includes three parts:

1. A questionnaire describing the occurrence of loco-regional morbidity in patients who has undergone breast conserving surgery with and without oncoplastic techniques.
2. Objective evaluation of shoulder and arm function and cosmesis before and after breast conserving surgery with and without oncoplastic techniques.
3. Long time follow-up of patients after breast conserving surgery without oncoplastic techniques.

Part 1

The questionnaire combines previous used and validated forms addressing shoulder and arm function, pain, sensibility, cosmesis and body image, and QoL. The questionnaire should be filled in preoperatively and 18 months after surgery. Patients included in the longtime follow-up study described below are asked to answer the same questionnaire, which includes questions about the following:

* Arm morbidity: Pain, sensibility, swelling, restriction of movements, force
* Quality of life (EORTC QLQ-C30 and QLQ-BR23)
* Comorbidity - Charlsons Comorbidity Index
* Body Image
* Physiotherapy Part 2

Cohort study with 18 months follow-up. Patients are evaluated at baseline before surgery and after 18 months with the following methods:

* Passive Range of movement (pROM). The passive motion of both shoulders are measured in supine position by use of a goniometer: flexion, extension, abduction, inner and outer rotation
* Constant Shoulder Score (CSS). Including active Range of movement (aROM) in flexion, abduction, rotation and strengths during shoulder abduction in upright standing position with the IsoForceControl dynamometer
* Sensibility recording
* Arm circumference
* Arm volume - simplified water displacement method
* Cosmetic outcome - using clinical photos of the breast region (frontal- and side view) and estimation of BRA (Breast Retraction Assessment) Re. part 1 and 2

Inclusion:

Patients, who are undergoing breast conserving surgery for invasive breast cancer or carcinoma in situ by one of the three breast surgical units at hospitals in Central Denmark Region (Viborg, Randers, and Aarhus). They will be divided in the two groups:

* BCS including oncoplastic surgical techniques
* BCS without oncoplastic surgical techniques

Exclusion:

* Patients who are unable to sign an informed consent form
* Patients above the age of 75 years and under the age of 18 years.
* Patients who have previously been operated in the same or the contralateral breast, shoulder or arm Part 3 The study performed by Husted Madsen et al. in 2003-4 included in all 395 patients. Surviving patients from this cohort are asked to e new evaluation of shoulder and arm function following the same procedure as described in Part 1 and 2.

Statistics:

Based on previous experience and statistical calculations estimated that the investigators need 495 to participate in the questionnaire (Part 1) and 220 patient for the objective evaluation (Part 2) Further details can be added If requested.

Ethics:

Patients included in part 1 and 2 will be contacted in the breast units after confirmation of the diagnosis and after decision about the treatment has been made. Before inclusion oral and written information about the study are given and the patient is asked to sign an informed consent form. For part 3 of these studies, patients receive a letter invitation and these patients are also asked to sign an informed consent form before entering the study.

There is only minor discomfort associated with the objective evaluation and no major complications or side effects are expected.

The protocol is submitted to The Local Research Ethics Committee for Central Region Denmark for approval.

ELIGIBILITY:
Inclusion Criteria:

* Invasive breast cancer or carcinoma in situ
* Breast conserving surgery including or without oncoplastic surgical techniques

Exclusion Criteria:

* Patients who are unable to sign an informed consent form
* Patients above the age og 75 and under the age of 18
* Patients who have previously been operated in the same or the contralateral breast, shoulder or arm

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients, who are undergoing breast conserving surgery (including or without oncoplastic surgical techniques) for invasive breast cancer or carcinoma in situ by one of the three breast surgical units in Central Denmark (Viborg, Randers and Aarhus).
  And surviving patients from the study by Husted Madsen et. al in 2003-4 ("Sentinel Node Biopsy and Breast Cancer - Aspects of introducing the method in Denmark") are invited to a new evaluation of shoulder and arm function.
Sampling Method: Non-Probability Sample
Enrollment: 408 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Shoulder function | before and 18 months after surgery
  By measuring passive and active range of movement (ROM) in the shoulder, measuring strength by a dynamometer (IsoForceControl). Estimating Constant Shoulder Score.

SECONDARY OUTCOMES:
Quality of life | 18 months
  Comparing EORTC QLQ-c30 and br23 before and 18 months after surgery.

OTHER OUTCOMES:
lymphoedema of the breast and arm | 18 months
  Estimating arm lympoedema by the water displacement method and breast lymphoedema by clinical evaluation.
Cosmetic results | 18 months
  Comparing cosmetic results by clinical evaluation and photos including breast retraction assessment (BRA)

CONTACTS AND LOCATIONS:
Overall Officials: Katrine R. Hauerslev, MD, Principal Investigator — University Hospital of Aarhus
Locations (1):
- Surgical department P, Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hauerslev KR, Overgaard J, Damsgaard TE, Hvid HM, Balling E, Fischer L, Christiansen P. Oncoplastic breast surgery versus conventional breast conserving surgery - a prospective follow-up study of subjective loco-regional late morbidity. Acta Oncol. 2021 Jun;60(6):750-759. doi: 10.1080/0284186X.2021.1900907. Epub 2021 Mar 31. PMID 33788646